CLINICAL TRIAL: NCT02407301
Title: Voluntary Cough Airflow Dynamics and True Vocal Fold Kinematics in Persons With Reduced True Vocal Fold Mobility
Brief Title: Cough in Reduced True Vocal Fold Mobility
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400733
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Unilateral Vocal Cord Paresis; Unilateral Vocal Cord Paralysis
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Laryngeal function in cough: cough airflow measure, vocal tasks, true vocal fold movement, spirometry test, and maximum expiratory pressure (MEP) assessment will be performed in this group.
  Interventions: Other: cough airflow measure; Other: vocal tasks; Other: true vocal fold movement; Other: spirometry test; Other: maximum expiratory pressure (MEP)

INTERVENTIONS:
Other: cough airflow measure — Participants will produce multiple voluntary coughs for cough airflow assessment.
  Other Names: cough airflow assessment
Other: vocal tasks — The assessment of glottal closure will be performed during phonation tasks.
  Other Names: phonation tasks
Other: true vocal fold movement — The true vocal fold (TVF) movement in cough will be observed and recorded during cough production.
  Other Names: TVF movement
Other: spirometry test — The lung function test will require the participant to perform deep inhalations and forceful exhalations into the flow head of the spirometer during spirometry test.
  Other Names: spirometry
Other: maximum expiratory pressure (MEP) — The assessment of maximum expiratory pressure will require forceful exhalations into a mouthpiece of a manometer during maximum expiratory pressure (MEP) assessment.
  Other Names: MEP

SUMMARY:
This project is a first attempt to assess cough airflow dynamics and true vocal fold (TVF) adduction and abduction angles during voluntary cough to examine the effects of changes in glottal closure due to reduced mobility of one true vocal fold. The hypothesis of this study is that the incomplete glottal closure due to reduced vocal fold mobility will result in changes in true vocal fold adductory and abductory angles during cough and will result in changes to voluntary cough airflow parameters. This study results will contribute to the existing knowledge of the laryngeal contribution to cough airflow dynamics.

DETAILED DESCRIPTION:
The study investigators will consecutively recruit 30 adults diagnosed with vocal fold insufficiency due to reduced mobility of one true vocal fold.

A questionnaire will be used to collect participants' information. Demographic information such as age, gender, race/ethnicity, height, weight, and a major complaint (dysphonia and/or dysphagia) and medical history information determining the eligibility for participation will be collected from the participant. Participant's medical and surgical history specifically related to the diagnosis and the etiology of reduced vocal fold mobility will be obtained from the participant's medical record.

Videolaryngoscopy will be performed as part of standard clinical care. Vocal fold image and cough airflow will be recorded simultaneously during voluntary cough production with the flexible endoscope in nasopharynx. A second part of the study will include spirometry and expiratory muscle strength assessments. Video images of the vocal fold movement during vowel phonation and cough production will be recorded and stored on a CD for later analysis. The cough airflow recordings will be displayed, stored, and analyzed using LabChart software for Windows.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 75 years.
2. Glottal insufficiency secondary to reduced TVF mobility confirmed with the endoscopic evaluation performed by an otolaryngologist.
3. The ability to provide informed consent.
4. No history of chronic obstructive pulmonary disease, lung cancer, and/or lung transplant.
5. No history of neurodegenerative disease such as Parkinson's disease, multiple sclerosis (MS), amyotrophic lateral sclerosis (ALS), or progressive supranuclear palsy (PSP), Alzheimer's disease, or dementia.

Exclusion Criteria:

1. Chest infection within one month prior to the study participation.
2. History of the adverse reaction associated with laryngoscopy.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will represent a population of patients with glottal insufficiency due to unilateral true vocal fold immobility.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Peak expiratory flow rate (PEFR) | baseline
  Maximum flow rate in expiratory phase, expressed in liters per second (L/s)
True vocal fold maximum abduction angles in inspiratory phase | baseline
  The TVF maximum abduction angles during cough inspiratory phase of cough will be expressed in degrees.
True vocal fold maximum abduction angles in expiratory phase | baseline
  True vocal fold maximum abduction angles in expiratory phase of cough will be expressed in degrees.
True vocal fold maximum adduction angles in compression phase | baseline
  True vocal fold maximum adduction angles in compression phase of cough will be expressed in degrees.
Peak expiratory flow rise time (PEFRT) | baseline
  Time to reach peak expiratory flow rate expressed in seconds
Cough volume acceleration (CVA) | baseline
  A ratio of peak expiratory flow rate and peak expiratory flow rise time expressed in L/s/s
Expiratory phase duration | baseline
  Duration of expiratory phase of cough expressed in seconds

SECONDARY OUTCOMES:
Peak expiratory flow | baseline
  Maximum flow rate during forced exhalation expressed in L/s
Maximum expiratory pressure | baseline
  Maximum expiratory pressure will be expressed in cmH2O.
Degree of glottal closure | baseline
  The degree of glottal closure will be assessed during phonation using glottic closure rating scale 1-6, 1=complete closure, 6=incomplete closure all along the vocal folds (Södersten et al., 1990).
Forced vital capacity (FVC) | baseline
  Maximum amount of air that can be exhaled with maximal speed and effort after maximum inhalation, expressed in L
Forced expired volume within 1 second (FEV1) | baseline
  Maximum amount of air exhaled forcefully within 1 second, expressed in L.
The ratio FEV1/FVC | baseline
  The percent (%) of forcefully exhaled air that can be exhaled during the first second of exhalation.

CONTACTS AND LOCATIONS:
Overall Officials: Karen W Hegland, Ph.D., Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida ENT Clinic, Gainesville, Florida
  - University of Florida Speech and Hearing Center, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Undecided